CLINICAL TRIAL: NCT04541095
Title: A Randomized, Multicenter, Controlled Clinical Trial to Assess Weight Gain of Preterm Infants Fed a New Infant Milk Formula Containing High Amounts of Beta-palmitate Versus a Standard Infant Milk Formula Containing Low Amounts of Beta-palmitate
Brief Title: Growth of Preterm Infants Fed a Infant Milk Formula Containing High Versus Low Amounts of Beta-palmitate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedali Riuniti Ancona (Other)
Collaborators: Istituto di Ricerca Pediatrica Città della Speranza (Unknown); Bunge Loders Croklaan (Industry)
Responsible Party: Principal Investigator, Virgilio Paolo Carnielli, The Director of Neonatology, Ospedali Riuniti Ancona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PG-1
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Weight Gain
Keywords: Growth; Preterm Infants; Beta-palmitate; Infant formula; Human milk
MeSH Terms: conditions — Weight Gain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EX_IMF group (Experimental): Infants will receive infants formula with large amounts of beta-palmitate (EX_IMF).
  Interventions: Other: EX_IMF
- ST_IMF group (Active Comparator): Infants will receive infants formula with low amounts of beta-palmitate (ST_IMF).
  Interventions: Other: ST_IMF
- HM group (No Intervention): Infants will receive human milk (HM).

INTERVENTIONS:
Other: EX_IMF — Infant formula with large amounts of beta-palmitate (about 60%).
  Arms: EX_IMF group
Other: ST_IMF — Infant formula with low amounts beta-palmitate (about 10%).
  Arms: ST_IMF group

SUMMARY:
The aim of this study is to assess weight gain of preterm infants (gestational age lower than 32 weeks) fed infant milk formula with about 60% beta-palmitate (EX_IMF) vs infant milk formula with similar macronutrient, mineral and fatty acid composition but lower amounts of beta-palmitate (ST_IMF). Own mother milk (OMM) fed infants will serve as reference group.

DETAILED DESCRIPTION:
A large number of low birth weight infants during their hospital stay experience poor growth and this has been linked to reduced neurodevelopment scores.

Several enriched infant milk formulas are available for preterm infants who cannot be fed human milk. The use of infant milk formulas (IMF) enriched with triglycerides similar to human milk lipids have shown to be associated with better fatty acid and mineral intestinal absorption.

In this multicenter, randomized, controlled clinical trial, preterm infants (gestational age lower than 32 weeks), who can not be fed human milk, will be randomized to receive IMF with high or low amounts of beta-palmitate (about 60% vs 10%, respectively). A non-randomized own human milk-fed group will be included as a reference. Patients will be on the study diet as soon as possible after birth and till 36 weeks of gestation. Neurodevelopment follow-up will be performed at 24 months corrected age.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 24 and 32 weeks of gestation at enrollment,
* birth weight greater than 750 grams,
* singleton or twin birth (no triplet or higher),
* fraction of inspired oxygen lower than 0.60 at enrollment,
* feasible enteral feeding,
* cardiovascular stable condition,
* informed consent form signed by at least one parent or legal guardian.

Exclusion Criteria:

* congenital malformations, genetic, metabolic and endocrine disorders,
* suspicious infection at enrollment,
* intrauterine growth restriction (<10th centile) at enrollment,
* maternal diabetes requiring insulin therapy,
* neonatal asphyxia.

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Weight gain | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Body weight will be daily measured by using an electronic balance (g/kg).

SECONDARY OUTCOMES:
Crying | For 1 consecutive day at 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Crying duration will be electronically recorded by a unidirectional microphone (hours/day).
Physical activity | For 1 consecutive day at 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before..
  The number of spontaneous movements per hour will be electronically measured by Kinect system.
Stooling pattern | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Stooling pattern will be reported by the parents according to on the Bristol stool form scale (consistency).
Stool biochemical composition - Total fatty acids | At 32 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Total fatty acids in the stool samples will be measured by gas chromatography (mg/g of dry feces).
Stool biochemical composition - Palmitic acid | At 32 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Palmitic acid in the stool samples will be measured by gas chromatography (mg/g of dry feces).
Stool biochemical composition - Calcium | At 32 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Fecal calcium will be measured by inductively coupled plasma emission spectrometry.
Stool biochemical composition - Phosphorus | At 32 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Fecal phosphorus will be measured by inductively coupled plasma emission spectrometry
Stool biochemical composition - Magnesium | At 32 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Fecal magnesium will be measured by inductively coupled plasma emission spectrometry.
Stool biochemical composition - Hydroxylic acids | At 32 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Fecal hydroxylic acids will be measured by high-resolution capillary chromatography
Infant formula intakes | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Cumulative infants formulas intakes (mL/kg).
Human milk intakes | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Cumulative human milk intakes (mL/kg).
Parenteral nutrition intakes - cumulative volume | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Cumulative parenteral nutrition intakes (mL/kg).
Parenteral nutrition intakes - amino acids | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Cumulative intravenous amino acid intakes (g/kg).
Parenteral nutrition intakes - glucose | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Cumulative intravenous glucose intakes (g/kg).
Parenteral nutrition intakes - lipids | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Cumulative intravenous lipid intakes (g/kg).
Parenteral nutrition duration | From birth to 36 weeks of gestational age or until discharge if this occurred before.
  Duration of parenteral nutrition (days)
Urinary dicarboxylic acid excretion | At 32 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Urinary dicarboxylic acids will be measured by gas chromatography-mass spectrometry (mmol/mol of creatinine).
Body weight | At 32, 34 and 36 weeks of gestational age or until discharge if this occurred before and then at 24 months of corrected age..
  Body weight will be measured by using an electronic balance (grams).
Total body length | At 32, 34 and 36 weeks of gestational age or until discharge if this occurred before and then at 24 months of corrected age.
  Total body length will be measured by using a stadiometer (cm).
Head circumference | At 32, 34 and 36 weeks of gestational age or until discharge if this occurred before and then at 24 months of corrected age.
  Head circumference will be measured by using a unstretchable tape (cm).
Blood biochemistry - Glycaemia | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Glucose concentrations in blood (mg/dL).
Blood biochemistry - Triglycerides | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Triglyceride concentrations in blood (mg/dL).
Blood biochemistry - Cholesterol | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Plasma cholesterol by gas chromatography-mass spectrometry (mg/dL).
Blood biochemistry - Phospholipids | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Plasma phospholipids by gas chromatography (mg/dL).
Blood biochemistry - Fatty acids | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Plasma total fatty acids by gas chromatography (mg/dL).
Blood biochemistry - Urea | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Urea concentrations in plasma (mg/dL).
Blood biochemistry - Bilirubin | At 7 and 42 days of postnatal age.
  Total and conjugated bilirubin concentrations (mg/dL).
Blood biochemistry - Electrolytes | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Na+, K+, Ca2+, Cl- and standard base excess (mmol/L).
Blood biochemistry - Calcium | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Calcium concentrations in blood (mg/dL).
Blood biochemistry - Phosphorus | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  phosphorus concentrations in blood (mg/dL).
Total body water | At 36 weeks of gestational age or until discharge if this occurred before.
  Total body water (% of body weight) will be measured by the deuterium dilution method.
Stool bifidobacteria | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Number of bifidobacteria per gram of feces will be measured by using fluorescent in situ hybridization.
Gastrointestinal problems | Daily from birth to 36 weeks of gestational age or until discharge if this occurred before.
  The incidence of gastrointestinal problems such as abdominal distension, gastric residuals, reflux and vomiting.
In-hospital death | Daily from birth to 36 weeks of gestational age or until discharge if this occurred before.
  The incidence of death during the hospital stay.
Complications of prematurity | Daily from birth to 36 weeks of gestational age or until discharge if this occurred before.
  The incidence of complications of prematurity such as respiratory distress syndrome (RDS), necrotizing enterocolitis (NEC), patent ductus arteriosus (PDA), intraventricular hemorrhage (IVH), retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), Periventricular Leukomalacia (PVL), sepsis, and cholestasis.
Neurodevelopmental assessment | At 24 months of corrected age.
  Neurodevelopment will be assessed by the Bayley test III.
Urinary urea | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Urea concentrations in urine (mg/dL).
Urinary calcium | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Calcium concentrations in urine (mg/dL).
Urinary phosphorus | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Phosphorus concentrations in urine (mg/dL).
Liver function tests | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Plasma alkaline phosphatase (ALP, IU/L), aspartate transaminase (AST, IU/L), alanine aminotransferase (ALT, IU/L) and gamma glutamyltranspeptidase concentrations (γ-GT, IU/L).
Parathyroid hormone | At 32, 34 and then at 36 weeks of gestational age or until discharge if this occurred before.
  Parathyroid hormone concentrations in blood (pg/mL).
Metabolic complications | Daily from birth to 36 weeks of gestational age or until discharge if this occurred before.
  hypo/hypernatremia, hypo/hyperkalemia, hypo/hyperchloremia, hypo/hypercalcemia, hypo/hyperparathyroidism, metabolic acidosis, hypo/hyperglycaemia, hypertriglyceridemia and elevated urea.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedali Riuniti di Ancona, Ancona
  - Istituto di Ricerca Città della Speranza, Padua

REFERENCES:
- [Background] Ehrenkranz RA, Younes N, Lemons JA, Fanaroff AA, Donovan EF, Wright LL, Katsikiotis V, Tyson JE, Oh W, Shankaran S, Bauer CR, Korones SB, Stoll BJ, Stevenson DK, Papile LA. Longitudinal growth of hospitalized very low birth weight infants. Pediatrics. 1999 Aug;104(2 Pt 1):280-9. doi: 10.1542/peds.104.2.280. PMID 10429008
- [Background] Hack M, Breslau N, Weissman B, Aram D, Klein N, Borawski E. Effect of very low birth weight and subnormal head size on cognitive abilities at school age. N Engl J Med. 1991 Jul 25;325(4):231-7. doi: 10.1056/NEJM199107253250403. PMID 2057024
- [Background] Innis SM, Dyer R, Nelson CM. Evidence that palmitic acid is absorbed as sn-2 monoacylglycerol from human milk by breast-fed infants. Lipids. 1994 Aug;29(8):541-5. doi: 10.1007/BF02536625. PMID 7990660
- [Background] Straarup EM, Lauritzen L, Faerk J, Hoy Deceased CE, Michaelsen KF. The stereospecific triacylglycerol structures and Fatty Acid profiles of human milk and infant formulas. J Pediatr Gastroenterol Nutr. 2006 Mar;42(3):293-9. doi: 10.1097/01.mpg.0000214155.51036.4f. PMID 16540799
- [Background] Carnielli VP, Luijendijk IH, Van Goudoever JB, Sulkers EJ, Boerlage AA, Degenhart HJ, Sauer PJ. Structural position and amount of palmitic acid in infant formulas: effects on fat, fatty acid, and mineral balance. J Pediatr Gastroenterol Nutr. 1996 Dec;23(5):553-60. doi: 10.1097/00005176-199612000-00007. PMID 8985844
- [Background] Carnielli VP, Luijendijk IH, van Goudoever JB, Sulkers EJ, Boerlage AA, Degenhart HJ, Sauer PJ. Feeding premature newborn infants palmitic acid in amounts and stereoisomeric position similar to that of human milk: effects on fat and mineral balance. Am J Clin Nutr. 1995 May;61(5):1037-42. doi: 10.1093/ajcn/61.4.1037. PMID 7733025
- [Background] Lucas A, Quinlan P, Abrams S, Ryan S, Meah S, Lucas PJ. Randomised controlled trial of a synthetic triglyceride milk formula for preterm infants. Arch Dis Child Fetal Neonatal Ed. 1997 Nov;77(3):F178-84. doi: 10.1136/fn.77.3.f178. PMID 9462186